CLINICAL TRIAL: NCT04027556
Title: Low-contrast Dose Liver CT Using Lean Body Weight, Low Monoenergetic Images and Deep Learning-based Reconstruction for Hepatocellular Carcinoma
Brief Title: Low-contrast Dose Liver CT Using Lean Body Weight Low Monoenergetic Images and Deep Learning-based Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: SNUH-2019-0344
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Hepatocellular; Body Weight
MeSH Terms: conditions — Carcinoma, Hepatocellular; Body Weight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 keV DLD images of the LBW-based low-dose group (Experimental): Low CT contrast media dose calculated based on lean body weight and low monoenergetic images of dual-energy CT with deep learning-based denoising
  Interventions: Other: low dose CT contrast media - lean body weight
- ADMIRE images of the standard-contrast dose group (Active Comparator): Standard CT contrast media dose calculated based on total body weight and conventional images with full model-based iterative reconstruction
  Interventions: Other: Standard dose CT contrast media

INTERVENTIONS:
Other: low dose CT contrast media - lean body weight — CT contrast media (iobitridol 350mgI/kg) is administrated at a dose of 450mgI/kg based on lean body weight.
  Arms: 50 keV DLD images of the LBW-based low-dose group
Other: Standard dose CT contrast media — CT contrast media (iobitridol 350mgI/kg) is administrated at a dose of 560mgI/kg based on total body weight.
  Arms: ADMIRE images of the standard-contrast dose group

SUMMARY:
This study aims to assess whether the acceptable image quality is achievable using low monoenergetic imaging of dual-energy CT with deep learning-based denoising, and low contrast media dose calculated based on lean body weight for the detection of hepatocellular carcinoma.

DETAILED DESCRIPTION:
The use of iodinated contrast media in CT is associated with an immediate hypersensitivity reaction in a dose-dependent manner. Therefore, it is important to reduce the contrast dose for CT exams in patients who are required repeated CT examinations, including patients with hepatocellular carcinoma (HCC). Low monoenergetic images of dual-energy CT can provide higher iodine contrast than conventional images, thus enabling reduction of contrast media. The high image noise in low monoenergetic images may be improved by using model-based IR techniques and deep learning-based denoising (DLD) algorithms. Besides, lean body weight (LBW)-based contrast dose determination can be another option to reduce contrast media dose compared with total body weight-based dose determination since the volumes of blood and liver are not strictly proportional to total body weight. Therefore, we surmised that 50 keV images reconstructed with DLD algorithms with reducing iodine load by 30% based on LBW could produce the comparable image quality and lesion conspicuity compared with standard iodine-dose 120kVp images.

In this single-center prospective, randomized clinical trial, we aimed to investigate the effectiveness of low-contrast dose CT using 50 keV and DLD technique compared with the standard contrast-dose protocol using model-based IR in patients at high risk of HCC.

ELIGIBILITY:
Inclusion Criteria:

* High risk group for developing HCC
* Scheduled contrast-enhanced CT for HCC diagnosis or surveillance

Exclusion Criteria:

* not a high risk group for developing HCC
* body mass index is equal to or larger than 30 kg/m^2
* suspected HCC > 5cm in diameter
* received locoregional treatment or surgery for HCC within 3 months
* congestive hepatopathy
* no venous access on forearm
* anticipated beam hardening artifact due to prosthesis
* relative/absolute contraindication of contrast-enhanced CT

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
HCC conspicuity | 6 months after complete enrollment
  qualitative scoring for focal lesion depiction on four-point scale (1: worst, 4: excellent, representative value is average score)

SECONDARY OUTCOMES:
Image noise | 12 months after complete enrollment
  qualitative scoring for image noise on four-point scale (1: worst, 4: excellent, representative value is average score)
Image contrast | 12 months after complete enrollment
  qualitative scoring for image contrast on four-point scale (1: worst, 4: excellent, representative value is average score)
Overall image quality | 6 months after complete enrollment
  qualitative scoring for image quality on four-point scale (1: worst, 4: excellent, representative value is average score)
Lesion detection | 12 months after complete enrollment
  assessment of focal liver lesion (HCC) on CT according to Liver Imaging Reporting and Data System (LI-RADS)
Hounsfield unit | 3 months after complete enrollment
  measurement of hounsfield unit in aorta, portal vein, liver parenchyma, and paraspinal muscles
Contrast media dose | 3 months after complete enrollment
  administered contrast media dose in each group
Radiation dose | 3 months after complete enrollment
  measured radiation dose in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No